CLINICAL TRIAL: NCT05220241
Title: Investigation of the Persistence of SARS-CoV-2 in the Olfactory Mucosa of Patients With Prolonged Symptoms of COVID-19 With Neurocognitive Complaints: a Prospective Cross-sectional Multicenter Case / Control Study (NEUROCOVID)
Brief Title: Investigation of the Persistence of SARS-CoV-2 in the Olfactory Mucosa of Patients With Prolonged Symptoms of COVID-19
Acronym: NEUROCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Hotel Dieu Hospital (Other); Institut Pasteur (Industry); Hôpital Lariboisière Fernand Widal (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MVT_2021_26
Record Dates: First submitted 2022-02-01; First posted 2022-02-02 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: SARS-CoV-2 Infection; Cognitive Disorder
MeSH Terms: conditions — COVID-19; Cognitive Dysfunction | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case : patient with 1st episode of COVID-19 and persistence of neurocognitive complaint (Other): Patient with a 1st episode of COVID-19 in the 12 months preceding inclusion and presenting persistence of neurocognitive complaint beyond 4 weeks
  Interventions: Biological: Nasopharyngeal swab for RT-PCR SARS-CoV-2
- Control : Patient with a 1st episode of COVID-19 cured and without neurocognitive complaint (Other): Patient with a cured 1st episode of COVID-19 (without persisting symptoms beyond 4 weeks) in the 12 months preceding inclusion and without neurocognitive complaint
  Interventions: Biological: Nasopharyngeal swab for RT-PCR SARS-CoV-2

INTERVENTIONS:
Biological: Nasopharyngeal swab for RT-PCR SARS-CoV-2 — 2 nasal swabs (one per nostril) of olfactory mucosa cells under local anesthesia for SARS-CoV-2 RT-PCR and pathological analysis
  Other Names: Blood sample for SARS-CoV-2 serology; MoCA (Control only); Ask the 3 questions from the Catherine Thomas-Antérion scale to search for a neurocognitive complaint (Control only)

SUMMARY:
NEUROCOVID is a prospective multicenter study comparing the proportion of patients with SARS-CoV-2 viral RNA at the level of the olfactory clefts in a group of cases compared to a group of controls as well as the correlations between the virological and cellular abnormalities observed in the olfactory mucosa and the severity of the clinical neurological profile

DETAILED DESCRIPTION:
More than 15% of people who developed COVID-19 would still have at least one symptom six months older. In France, this would concern several hundred thousand people. The societal consequences are important. The symptoms are very polymorphic; they evolve in a fluctuating fashion and persist for several months. Neurological symptoms are often in the foreground and include different symptoms, among which:

* Cognitive disorders (psychic slowing down, lack of clarity in thought, difficulty in remembering certain facts, difficulty in performing double tasks, difficulty in finding words).
* Sensory disturbances such as burning or tingling with or without root topography, dizziness.
* Neurovegetative manifestations: sudden tachycardia, palpitations, vasomotor disorders, excessive sweating, digestive disorders or post prandial malaise, feelings of malaise (lipothymia with or without hypotension), dyspnea or a feeling of dyspnea, urinary disorders
* Sleep disorders (insomnia, sleep fragmentation, nightmares or hypersomnia)
* Tension type headaches.

The mechanisms explaining the occurrence of these symptoms are still debated. An important result is the recent demonstration by the UK's National Statistics Office that people with "long COVID" may, for some, remain carriers of the SARS-CoV-2 virus for several months. So far, viral persistence has only been demonstrated in a few specific cases of immunocompromised people, almost all of them having been hospitalized.

Recently, in a pilot study conducted jointly by the Institut Pasteur and AP-HP, we demonstrated that viral RNA could be found in immunocompetent patients with prolonged neurological symptoms after COVID-19 (Melo et al 2021). This study concerned 4 patients explored by micro-brushing the mucous membrane of the olfactory cracks under local anesthesia more than 4 months after the initial COVID-19. In all patients, SARS-CoV-2 RNA persisted in significant amounts.

Although this demonstration currently only concerns a small number of people, this study provides evidence that the virus can remain hidden in the olfactory cracks (a tissue that is part of the nervous system), including in people with PCR nasopharyngeal and / or SARS-CoV-2 serology become negative. This persistence of the virus after a so-called "acute" infection is not unique. In EBOLA virus disease, some people have been shown to keep the virus in their semen for several months.

It is now necessary to determine whether this persistence is specific to long COVID, what are the mechanisms and the consequences of this persistence of the virus.

One of the hypotheses is that the virus would persist in endothelial cells and / or support cells. Intermittent reactivation of the virus would lead to intermittent inflammation, secretion of pro-inflammatory cytokines, activation of coagulation and innate immunity cells (monocytes, mast cells, astrocytes, cerebral glial cells) or adaptive This activation could be due to origin of possible micro-thrombosis responsible for a decrease in the oxygen supply in the tissues. This tissue hypoxia could cause the intermittent "brain fog" complained about by patients and the cerebral hypo-metabolisms seen on CT scans. The virus could infect other cells as well, and the issue of direct infection of neurons remains unresolved.

In this study, we want to assess whether viral persistence is specific to patients with prolonged symptoms following COVID-19, to assess whether the presence of SARS-CoV-2 RNA is correlated with the ability of the virus to replicate, study the cellular abnormalities associated with the presence of viruses, and correlate the observed cellular and virological abnormalities with the clinical profile of patients.

We are interested in central neurological disorders, in particular cognitive disorders, because they are often in the foreground, and they are by far the most disabling symptoms for patients.

ELIGIBILITY:
Inclusion Criteria:

Common to cases and controls:

* Age ≥ 18 years old and <60 years old
* Good oral and written command of French
* Level of education ≥ 7 years of schooling
* Initial episode of COVID-19 within 2 to 12 months
* Symptomatic initial episode of COVID-19
* Initial symptoms not explained by another diagnosis
* Initial episode documented by RT-PCR positive for SARS-CoV-2 and / or positive antigen test and / or positive serology (in the absence of vaccination)
* Express consent to participate in the study
* Affiliate or beneficiary of a social security scheme

Case group:

* Presence of at least one of the initial symptoms beyond 4 weeks following the onset of the acute phase of the disease
* Prolonged symptoms not explained by another diagnosis with no known link to COVID-19
* Neurocognitive complaint (s) previously objectified by a neurologist and after completion of a neuro-psychological assessment
* Impact of neurocognitive disorders on daily life authenticated by a Glasgow outcome scale extended ≤ 7 (see appendix 1)
* Evolution of complaints for 2 to 12 months compared to the date of their first appearance

Exclusion Criteria:

Exclusion criteria common to cases and controls:

* Person benefiting from a legal protection measure
* Pregnant or breastfeeding woman
* At least one neurological pathology among:

  * encephalopathy
  * encephalitis
  * severe neurological form of the initial episode of COVID-19
  * neurodegenerative disease
* History of stroke
* Serious psychiatric history
* Known nasal sinus pathology
* Hemostatic disorder
* Taking aspirin in the 15 days preceding the sample
* Treatment with anticoagulants
* Known allergy to lidocaine

Secondary exclusion criteria for controls:

- Positive SARS-CoV-2 RT-PCR on nasopharyngeal sample on the day of inclusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Presence of SARS-CoV-2 RNA in the olfactory mucosa | Inclusion
  Comparison of the presence of SARS-CoV-2 RNA in the olfactory mucosa between cases and controls

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Veyrat, Dr, Principal Investigator — Hôpital Fondation A. de Rothschild
Locations (2):
- France (2):
  - Hôpital Lariboisière-Fernand-Widal, Paris
  - Hôpital Fondation A. de Rothschild, Paris